CLINICAL TRIAL: NCT00830063
Title: A PHASE 3 RANDOMIZED, DOUBLE BLIND PLACEBO AND NAPROXEN CONTROLLED MULTICENTER STUDY OF THE ANALGESIC EFFICACY AND SAFETY OF TANEZUMAB IN PATIENTS WITH OSTEOARTHRITIS OF THE KNEE
Brief Title: Tanezumab In Osteoarthritis Of The Knee (2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A4091015; P3 OA KNEE NSAID POPULATION (Other: Alias Study Number)
Record Dates: First submitted 2009-01-23; First posted 2009-01-27 (Estimated); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Arthritis; Osteoarthritis
Keywords: monoclonal antibody; RN624; PF-04383119; nerve growth factor; anti-nerve growth factor; OA; pain
MeSH Terms: conditions — Arthritis; Osteoarthritis; Hereditary Sensory and Autonomic Neuropathies; Pain | interventions — tanezumab; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental)
  Interventions: Biological: tanezumab 10 mg
- 2 (Experimental)
  Interventions: Biological: tanezumab 5 mg
- 3 (Active Comparator)
  Interventions: Drug: naproxen
- 4 (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Biological: tanezumab 10 mg — tanezumab 10 mg one dose at weeks 0 and 8
  Arms: 1
Biological: tanezumab 5 mg — tanezumab 5 mg one dose at weeks 0 and 8
  Arms: 2
Drug: naproxen — naproxen 1000 mg daily for 16 weeks
  Arms: 3
Other: placebo — placebo to match tanezumab and naproxen dosing
  Arms: 4

SUMMARY:
The purpose of this study is to test the efficacy and safety of 2 doses of tanezumab compared with naproxen and placebo in patients with osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee according to Kellgren-Lawrence x-ray grade of 2

Exclusion Criteria:

* Pregnancy or intent to become pregnant
* BMI greater than 39
* other severe pain, significant cardiac, neurologic or cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 832 (Actual)
Dates: Start 2009-05-05 (Actual); Primary Completion 2010-05-17 (Actual); Study Completion 2010-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (94):
- United States (94):
  - Anniston Medical Clinic, PC, Anniston, Alabama
  - Pinnaccle Research Group, LLC, Anniston, Alabama
  - Clinical Research Advantage, Inc. / Mesa Family Medical Center, PC, Mesa, Arizona
  - Arizona Arthritis & Rheumatology Associates, P.C., Paradise Valley, Arizona
  - Pivotal Research Centers, Peoria, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Arizona Arthritis & Rheumatology Associates, P.C., Phoenix, Arizona
  - University of Arizona - Arizona Arthritis Center, Tucson, Arizona
  - University of Arizona, Tucson, Arizona
  - St. Joseph's Mercy Clinic, Hot Springs, Arkansas
  - Osteoporosis Medical Center, Beverly Hills, California
  - Valley Research, Fresno, California
  - Talbert Medical Group, Huntington Beach, California
  - UC Davis Medical Center, Sacramento, California
  - Lawrence P McAdam, MD / A Medical Corporation, Thousand Oaks, California
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Javed Rheumatology Associates, Inc., Newark, Delaware
  - Innovative Research of West Florida, Inc, Clearwater, Florida
  - Tampa Bay Medical Research, Inc., Clearwater, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Adult Medicine Specialists, Longwood, Florida
  - Genesis Research International, Longwood, Florida
  - Kendall South Medical Center, Inc, Miami, Florida
  - The Arthritis Center, Palm Harbor, Florida
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - Progressive Medical Research, Port Orange, Florida
  - West Broward Rheumatology Associates, Inc., Tamarac, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Arthritis and Rheumatology of Georgia, Atlanta, Georgia
  - Jeffrey D. Lieberman, MD, Decatur, Georgia
  - Marietta Rheumatology, Marietta, Georgia
  - Physician Pain Care, Woodstock, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - North Georgia Internal Medicine, Woodstock, Georgia
  - Sonora Clinical Research, Boise, Idaho
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Koch Family Practice, Morton, Illinois
  - Illinois Bone and Joint Institute, LLC, Morton Grove, Illinois
  - The Arthritis Center, Springfield, Illinois
  - Northwest Indiana Center for Clinical Research, Valparaiso, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Integrated Clinical Trial Services, Inc., West Des Moines, Iowa
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - David H. Neustadt, PSC, Louisville, Kentucky
  - Stanocola Medical Center, Baton Rouge, Louisiana
  - Maine Research Associates, Auburn, Maine
  - Arthritis and Osteoporosis Center of Maryland, Frederick, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Shores Rheumatology, P.C., Saint Clair Shores, Michigan
  - MAPS Applied Research Center, Inc, Edina, Minnesota
  - Medical Advanced Pain Specialists, Edina, Minnesota
  - Mercy Health Research, St Louis, Missouri
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Clinical Research Consortium, Las Vegas, Nevada
  - Mirkil Medical, Las Vegas, Nevada
  - G. Timothy Kelly, MD, Las Vegas, Nevada
  - Michael Clifford, MD, Las Vegas, Nevada
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - New Mexico Clinical Research & Osteoporosis Center, Incorporated, Albuquerque, New Mexico
  - The Medical Research Network, LLC, New York, New York
  - AAIR Research Center, Rochester, New York
  - Andrew J. Porges, MD, PC, Roslyn, New York
  - Carolina Bone and Joint, PA, Charlotte, North Carolina
  - Pharmquest, Greensboro, North Carolina
  - Odyssey Research, Fargo, North Dakota
  - Plains Medical Clinic, LLC, Fargo, North Dakota
  - Hightop Medical Research Center, Cincinnati, Ohio
  - Hilltop Physicians Inc / Hightop Medical Research Center, Cincinnati, Ohio
  - Southwest Rheumatology and Research Group, LLC, Middleburg Heights, Ohio
  - Pharmacotherapy Research Associates Incorporated, Zanesville, Ohio
  - Health Research Institute, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading, LLP, West Reading, Pennsylvania
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Appalachian Medical Research, Inc, Johnson City, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Capitol Medical Clinic, Austin, Texas
  - Office of Walter F Chase, MD, PA, Austin, Texas
  - North Texas Joint Care, PA, Dallas, Texas
  - Asif Cochinwala, MD, PA, Houston, Texas
  - Pioneer Research Solutions, Inc, Houston, Texas
  - Radiant Research San Antonio Northeast, San Antonio, Texas
  - Diagnostic Research Group, San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - South Texas Radiology Group, San Antonio, Texas
  - Aspen Clinical Research, LLC, Orem, Utah
  - National Clinical Research - Norfolk, Inc., Norfolk, Virginia
  - Arthritis and Rheumatic Diseases, Portsmouth, Virginia
  - Clinical Trials Northwest, Yakima, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Brown MT, Cornblath DR, Koltzenburg M, Gorson KC, Hickman A, Pixton GC, Gaitonde P, Viktrup L, West CR. Peripheral Nerve Safety of Nerve Growth Factor Inhibition by Tanezumab: Pooled Analyses of Phase III Clinical Studies in Over 5000 Patients with Osteoarthritis. Clin Drug Investig. 2023 Jul;43(7):551-563. doi: 10.1007/s40261-023-01286-3. Epub 2023 Jul 18. PMID 37460782
- [Derived] Tive L, Bello AE, Radin D, Schnitzer TJ, Nguyen H, Brown MT, West CR. Pooled analysis of tanezumab efficacy and safety with subgroup analyses of phase III clinical trials in patients with osteoarthritis pain of the knee or hip. J Pain Res. 2019 Mar 19;12:975-995. doi: 10.2147/JPR.S191297. eCollection 2019. PMID 30936738
- [Derived] Ekman EF, Gimbel JS, Bello AE, Smith MD, Keller DS, Annis KM, Brown MT, West CR, Verburg KM. Efficacy and safety of intravenous tanezumab for the symptomatic treatment of osteoarthritis: 2 randomized controlled trials versus naproxen. J Rheumatol. 2014 Nov;41(11):2249-59. doi: 10.3899/jrheum.131294. Epub 2014 Oct 1. PMID 25274899

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo matched to tanezumab (RN624 or PF-04383119) intravenous (IV) infusion at Day 1 and Week 8, and placebo matched to naproxen tablet orally twice daily (BID) from Day 1 to Week 16.
- Tanezumab 5 mg + Placebo: Participants received tanezumab (RN624 or PF-04383119) 5 milligram (mg) IV infusion at Day 1 and Week 8, and placebo matched to naproxen tablet orally twice daily from Day 1 to Week 16.
- Tanezumab 10 mg + Placebo: Participants received tanezumab (RN624 or PF-04383119) 10 mg IV infusion at Day 1 and Week 8, and placebo matched to naproxen tablet orally twice daily from Day 1 to Week 16.
- Naproxen + Placebo: Participants received naproxen 500 mg tablet orally twice daily from Day 1 to Week 16 and placebo matched to tanezumab (RN624 or PF-04383119) IV infusion at Day 1 and Week 8.
Period: Overall Study
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Started | 208 | 208 | 208 | 208
Treated | 208 | 206 | 208 | 206
Completed | 8 | 16 | 10 | 13
Not Completed | 200 | 192 | 198 | 195
Not completed — Adverse Event | 7 | 13 | 16 | 13
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 1
Not completed — Preferred Time Entry in Extension Study | 119 | 139 | 127 | 126
Not completed — Lack of Efficacy | 51 | 23 | 25 | 32
Not completed — Other | 5 | 5 | 8 | 6
Not completed — Withdrawal by Subject | 16 | 10 | 16 | 13
Not completed — Protocol Violation | 1 | 0 | 3 | 2
Not completed — Randomized But Not Treated | 0 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all randomized participants who received at least 1 dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo | Total
Number analyzed (Participants) | 208 | 206 | 208 | 206 | 828
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (10.1) | 61.1 (10.1) | 61.1 (10.3) | 61.4 (10) | 61.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 122 | 128 | 129 | 499
  Male | 88 | 84 | 80 | 77 | 329

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale at Week 16: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms in participants with osteoarthritis of knee. WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in the index knee during past 48 hours. It is calculated as mean of the scores from 5 individual questions scored on a numerical rating scale of 0 (minimum pain) to 10 (maximum pain), where higher scores indicate more pain. An overall possible WOMAC pain subscale score range is of 0 (minimum pain) to 10 (maximum pain), where higher scores indicate more pain.
Time Frame: Baseline (Day 1), Week 16
Population: Modified ITT (mITT): All participants who received at least 1 dose of the study drug, except those with concerns about data integrity at 1 of the study centers. BOCF method was used to impute missing values. Here "Overall number of participants analyzed (N)" signifies the participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 199 | 202 | 202 | 200
units on a scale
  Baseline | 7.21 (1.43) | 7.30 (1.47) | 7.25 (1.41) | 7.18 (1.37)
  Change at Week 16 | -2.23 (2.56) | -3.55 (2.84) | -3.27 (2.81) | -2.82 (2.54)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg + Placebo; Least square (LS) mean was estimated from the corresponding analysis of covariance (ANCOVA) model. ANCOVA model included treatment as main effects, baseline value, and study site as a random effect. 95 percent (%) confidence interval (CI) was calculated on LS mean difference; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS Mean difference = -1.24, 95% CI 2-sided [-1.76 to -0.72], Standard Error of Mean 0.26
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg + Placebo; LS mean was estimated from the corresponding ANCOVA model. ANCOVA model included treatment as main effects, baseline value, and study site as a random effect. 95% CI was calculated on LS mean difference; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.00, 95% CI 2-sided [-1.52 to -0.49], Standard Error of Mean 0.26
Statistical Analysis 3: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.007, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.72, 95% CI 2-sided [-1.23 to -0.20], Standard Error of Mean 0.26
Statistical Analysis 4: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.068, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.48, 95% CI 2-sided [-0.99 to 0.03], Standard Error of Mean 0.26

2. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale at Week 16: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms in participants with osteoarthritis of knee. WOMAC physical function subscale is a 17-item questionnaire used to assess the degree of difficulty experienced due to osteoarthritis in index knee joint during past 48 hours. It is calculated as mean of the scores from 17 individual questions scored on a numerical rating scale of 0 (minimum difficulty) to 10 (maximum difficulty), where higher scores indicate more difficulty. An overall possible WOMAC physical function subscale score range is of 0 (minimum difficulty) to 10 (maximum difficulty), where higher scores indicate worse function. Physical function refers to participant's ability to move around and perform usual activities of daily living.
Time Frame: Baseline, Week 16
Population: mITT population included all participants who received at least 1 dose of the study drug, except those with concerns about data integrity at 1 of the study centers. BOCF method was used to impute missing values. Here 'N' signifies the participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 198 | 202 | 201 | 200
units on a scale
  Baseline | 6.85 (1.56) | 6.86 (1.71) | 6.86 (1.50) | 6.86 (1.57)
  Change at Week 16 | -1.88 (2.29) | -3.18 (2.64) | -2.91 (2.59) | -2.42 (2.40)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.25, 95% CI 2-sided [-1.73 to -0.77], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.03, 95% CI 2-sided [-1.51 to -0.55], Standard Error of Mean 0.24
Statistical Analysis 3: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.76, 95% CI 2-sided [-1.24 to -0.28], Standard Error of Mean 0.24
Statistical Analysis 4: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.030, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.53, 95% CI 2-sided [-1.01 to -0.05], Standard Error of Mean 0.24

3. Primary Outcome: Change From Baseline in Patient Global Assessment of Osteoarthritis at Week 16: Baseline Observation Carried Forward (BOCF)
Description: Participants answered: "Considering all the ways the osteoarthritis in your index knee affects you, how are you doing today?" Participants responded on the scale ranging from 1 (minimum affected) to 5 (maximum affected), where 1= very good, 2= good, 3= fair, 4= poor and 5= very poor. Higher scores indicate worse condition.
Time Frame: Baseline, Week 16
Population: mITT population included all participants who received at least 1 dose of the study drug, except those with concerns about data integrity at 1 of the study centers. BOCF method was used to impute missing values. Here, 'N' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 198 | 201 | 202 | 200
units on a scale
  Baseline | 3.41 (0.61) | 3.41 (0.59) | 3.39 (0.55) | 3.44 (0.62)
  Change at Week 16 | -0.53 (0.83) | -0.87 (1.02) | -0.74 (0.88) | -0.70 (0.97)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.33, 95% CI 2-sided [-0.50 to -0.16], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.014, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.21, 95% CI 2-sided [-0.39 to -0.04], Standard Error of Mean 0.09
Statistical Analysis 3: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.026, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.19, 95% CI 2-sided [-0.36 to -0.02], Standard Error of Mean 0.09
Statistical Analysis 4: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.349, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.08, 95% CI 2-sided [-0.25 to 0.09], Standard Error of Mean 0.09

4. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale at Week 2, 4, 8 and 12: Baseline Observation Carried Forward (BOCF)
Description: as for outcome 1
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 199 | 202 | 202 | 200
units on a scale
  Change at Week 2 | -2.34 (2.26) | -2.61 (2.58) | -2.95 (2.53) | -3.12 (2.37)
  Change at Week 4 | -2.36 (2.31) | -3.59 (2.52) | -3.99 (2.64) | -3.28 (2.41)
  Change at Week 8 | -2.35 (2.35) | -3.63 (2.61) | -3.89 (2.77) | -3.13 (2.57)
  Change at Week 12 | -2.24 (2.56) | -3.89 (2.83) | -3.65 (2.92) | -2.98 (2.65)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg + Placebo; Week 2: LS mean was estimated from the corresponding ANCOVA model. ANCOVA model included treatment as main effects, baseline value, and study site as a random effect. 95% CI was calculated on LS mean difference; Test type: Superiority or Other; p = 0.355, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.22, 95% CI 2-sided [-0.69 to 0.25], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.017, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.57, 95% CI 2-sided [-1.04 to -0.10], Standard Error of Mean 0.24
Statistical Analysis 3: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.020, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = 0.56, 95% CI 2-sided [0.09 to 1.03], Standard Error of Mean 0.24
Statistical Analysis 4: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.388, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = 0.21, 95% CI 2-sided [-0.26 to 0.67], Standard Error of Mean 0.24
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 5 mg + Placebo; Week 4: LS mean was estimated from the corresponding ANCOVA model. ANCOVA model included treatment as main effects, baseline value, and study site as a random effect. 95% CI was calculated on LS mean difference; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.18, 95% CI 2-sided [-1.65 to -0.70], Standard Error of Mean 0.24
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.60, 95% CI 2-sided [-2.07 to -1.13], Standard Error of Mean 0.24
Statistical Analysis 7: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.274, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.26, 95% CI 2-sided [-0.73 to 0.21], Standard Error of Mean 0.24
Statistical Analysis 8: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.004, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.69, 95% CI 2-sided [-1.16 to -0.22], Standard Error of Mean 0.24
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 5 mg + Placebo; Week 8: LS mean was estimated from the corresponding ANCOVA model. ANCOVA model included treatment as main effects, baseline value, and study site as a random effect. 95% CI was calculated on LS mean difference; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.25, 95% CI 2-sided [-1.74 to -0.75], Standard Error of Mean 0.25
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.50, 95% CI 2-sided [-2.00 to -1.01], Standard Error of Mean 0.25
Statistical Analysis 11: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p = 0.051, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.49, 95% CI 2-sided [-0.99 to 0.00], Standard Error of Mean 0.25
Statistical Analysis 12: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; Slope = -0.75, 95% CI 2-sided [-1.24 to -0.25], Standard Error of Mean 0.25
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 5 mg + Placebo; Week 12: LS mean was estimated from the corresponding ANCOVA model. ANCOVA model included treatment as main effects, baseline value, and study site as a random effect. 95% CI was calculated on LS mean difference; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.59, 95% CI 2-sided [-2.12 to -1.07], Standard Error of Mean 0.27
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.37, 95% CI 2-sided [-1.90 to -0.85], Standard Error of Mean 0.27
Statistical Analysis 15: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.89, 95% CI 2-sided [-1.42 to -0.37], Standard Error of Mean 0.27
Statistical Analysis 16: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.012, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.67, 95% CI 2-sided [-1.19 to -0.15], Standard Error of Mean 0.27

5. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale at Week 2, 4, 8 and 12: Last Observation Carried Forward (LOCF)
Description: as for outcome 1
Time Frame: Baseline, Week 2, 4, 8, 12
Population: mITT population included all participants who received at least 1 dose of the study drug, except those with concerns about data integrity at 1 of the study centers. LOCF method was used to impute missing values. Here, 'N' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 199 | 202 | 202 | 200
units on a scale
  Baseline | 7.21 (1.43) | 7.30 (1.47) | 7.25 (1.41) | 7.18 (1.37)
  Change at Week 2 | -2.34 (2.26) | -2.61 (2.58) | -2.95 (2.53) | -3.12 (2.37)
  Change at Week 4 | -2.53 (2.32) | -3.58 (2.56) | -4.14 (2.51) | -3.32 (2.39)
  Change at Week 8 | -2.62 (2.35) | -3.73 (2.60) | -4.24 (2.53) | -3.26 (2.52)
  Change at Week 12 | -2.80 (2.50) | -4.07 (2.72) | -4.21 (2.56) | -3.34 (2.58)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.355, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS Mean difference = -0.22, 95% CI 2-sided [-0.69 to 0.25], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.017, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.57, 95% CI 2-sided [-1.04 to -0.10], Standard Error of Mean 0.24
Statistical Analysis 3: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.020, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = 0.56, 95% CI 2-sided [0.09 to 1.03], Standard Error of Mean 0.24
Statistical Analysis 4: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.388, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = 0.21, 95% CI 2-sided [-0.26 to 0.67], Standard Error of Mean 0.24
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.98, 95% CI 2-sided [-1.45 to -0.52], Standard Error of Mean 0.24
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.56, 95% CI 2-sided [-2.02 to -1.10], Standard Error of Mean 0.24
Statistical Analysis 7: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.361, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.22, 95% CI 2-sided [-0.68 to 0.25], Standard Error of Mean 0.24
Statistical Analysis 8: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.79, 95% CI 2-sided [-1.25 to -0.33], Standard Error of Mean 0.23
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.06, 95% CI 2-sided [-1.54 to -0.59], Standard Error of Mean 0.24
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.57, 95% CI 2-sided [-2.04 to -1.09], Standard Error of Mean 0.24
Statistical Analysis 11: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p = 0.063, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.45, 95% CI 2-sided [-0.93 to 0.02], Standard Error of Mean 0.24
Statistical Analysis 12: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.96, 95% CI 2-sided [-1.43 to -0.48], Standard Error of Mean 0.24
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.20, 95% CI 2-sided [-1.70 to -0.71], Standard Error of Mean 0.25
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.35, 95% CI 2-sided [-1.85 to -0.86], Standard Error of Mean 0.25
Statistical Analysis 15: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.006, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.70, 95% CI 2-sided [-1.19 to -0.21], Standard Error of Mean 0.25
Statistical Analysis 16: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.85, 95% CI 2-sided [-1.34 to -0.36], Standard Error of Mean 0.25

6. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale at Week 2, 4, 8 and 12: Baseline Observation Carried Forward (BOCF)
Description: as for outcome 2
Time Frame: Baseline, Week 2, 4, 8, 12
Population: mITT population included all participants who received at least 1 dose of the study drug, except those with concerns about data integrity at 1 of the study centers. BOCF method was used to impute missing values. Here, 'N' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 198 | 202 | 201 | 200
units on a scale
  Change at Week 2 | -1.92 (2.09) | -2.44 (2.48) | -2.80 (2.35) | -2.66 (2.40)
  Change at Week 4 | -1.92 (2.19) | -3.07 (2.47) | -3.63 (2.46) | -2.90 (2.38)
  Change at Week 8 | -1.96 (2.14) | -3.18 (2.47) | -3.50 (2.57) | -2.70 (2.52)
  Change at Week 12 | -1.93 (2.28) | -3.46 (2.70) | -3.32 (2.72) | -2.66 (2.53)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.355, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.22, 95% CI 2-sided [-0.69 to 0.25], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.017, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.57, 95% CI 2-sided [-1.04 to -0.10], Standard Error of Mean 0.24
Statistical Analysis 3: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.020, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = 0.56, 95% CI 2-sided [0.09 to 1.03], Standard Error of Mean 0.24
Statistical Analysis 4: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.388, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = 0.21, 95% CI 2-sided [-0.26 to 0.67], Standard Error of Mean 0.24
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.18, 95% CI 2-sided [-1.65 to -0.70], Standard Error of Mean 0.24
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.60, 95% CI 2-sided [-2.07 to -1.13], Standard Error of Mean 0.24
Statistical Analysis 7: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.274, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.26, 95% CI 2-sided [-0.73 to 0.21], Standard Error of Mean 0.24
Statistical Analysis 8: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.004, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.69, 95% CI 2-sided [-1.16 to -0.22], Standard Error of Mean 0.24
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.25, 95% CI 2-sided [-1.74 to -0.75], Standard Error of Mean 0.25
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.50, 95% CI 2-sided [-2.00 to -1.01], Standard Error of Mean 0.25
Statistical Analysis 11: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p = 0.051, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.49, 95% CI 2-sided [-0.99 to 0.00], Standard Error of Mean 0.25
Statistical Analysis 12: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.75, 95% CI 2-sided [-1.24 to -0.25], Standard Error of Mean 0.25
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; -1.59 = -1.59, 95% CI 2-sided [-2.12 to -1.07], Standard Error of Mean 0.27
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.37, 95% CI 2-sided [-1.90 to -0.85], Standard Error of Mean 0.27
Statistical Analysis 15: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.89, 95% CI 2-sided [-1.42 to -0.37], Standard Error of Mean 0.27
Statistical Analysis 16: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.012, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.67, 95% CI 2-sided [-1.19 to -0.15], Standard Error of Mean 0.27

7. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale at Week 2, 4, 8 and 12: Last Observation Carried Forward (LOCF)
Description: as for outcome 2
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 198 | 202 | 201 | 200
units on a scale
  Baseline | 6.85 (1.56) | 6.86 (1.71) | 6.86 (1.50) | 6.86 (1.57)
  Change at Week 2 | -1.92 (2.09) | -2.44 (2.48) | -2.80 (2.35) | -2.66 (2.40)
  Change at Week 4 | -2.02 (2.23) | -3.07 (2.54) | -3.73 (2.40) | -2.93 (2.37)
  Change at Week 8 | -2.13 (2.22) | -3.27 (2.50) | -3.77 (2.45) | -2.83 (2.51)
  Change at Week 12 | -2.31 (2.35) | -3.61 (2.67) | -3.79 (2.51) | -2.95 (2.52)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.026, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.51, 95% CI 2-sided [-0.96 to -0.06], Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.87, 95% CI 2-sided [-1.32 to -0.43], Standard Error of Mean 0.23
Statistical Analysis 3: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.333, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = 0.22, 95% CI 2-sided [-0.23 to 0.67], Standard Error of Mean 0.23
Statistical Analysis 4: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.527, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.14, 95% CI 2-sided [-0.59 to 0.30], Standard Error of Mean 0.23
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.03, 95% CI 2-sided [-1.48 to -0.57], Standard Error of Mean 0.23
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.71, 95% CI 2-sided [-2.16 to -1.25], Standard Error of Mean 0.23
Statistical Analysis 7: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.574, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.13, 95% CI 2-sided [-0.58 to 0.32], Standard Error of Mean 0.23
Statistical Analysis 8: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.81, 95% CI 2-sided [-1.26 to -0.36], Standard Error of Mean 0.23
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.13, 95% CI 2-sided [-1.60 to -0.67], Standard Error of Mean 0.24
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.64, 95% CI 2-sided [-2.10 to -1.17], Standard Error of Mean 0.24
Statistical Analysis 11: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p = 0.055, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.45, 95% CI 2-sided [-0.92 to 0.01], Standard Error of Mean 0.24
Statistical Analysis 12: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.96, 95% CI 2-sided [-1.42 to -0.49], Standard Error of Mean 0.24
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.27, 95% CI 2-sided [-1.75 to -0.79], Standard Error of Mean 0.24
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -1.47, 95% CI 2-sided [-1.95 to -0.99], Standard Error of Mean 0.24
Statistical Analysis 15: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.006, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.67, 95% CI 2-sided [-1.15 to -0.19], Standard Error of Mean 0.24
Statistical Analysis 16: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.87, 95% CI 2-sided [-1.34 to -0.39], Standard Error of Mean 0.24

8. Secondary Outcome: Change From Baseline in Patient Global Assessment of Osteoarthritis at Week 2, 4, 8 and 12: Baseline Observation Carried Forward (BOCF)
Description: as for outcome 3
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 198 | 201 | 202 | 200
units on a scale
  Change at Week 2 | -0.53 (0.78) | -0.69 (0.91) | -0.68 (0.90) | -0.89 (0.94)
  Change at Week 4 | -0.52 (0.75) | -1.02 (0.98) | -1.07 (0.90) | -0.89 (0.85)
  Change at Week 8 | -0.52 (0.81) | -0.95 (0.97) | -0.96 (0.95) | -0.77 (0.96)
  Change at Week 12 | -0.53 (0.74) | -0.98 (1.00) | -0.83 (0.94) | -0.73 (0.87)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.045, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.16, 95% CI 2-sided [-0.32 to -0.00], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.030, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.18, 95% CI 2-sided [-0.33 to -0.02], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.027, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = 0.18, 95% CI 2-sided [0.02 to 0.34], Standard Error of Mean 0.08
Statistical Analysis 4: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.040, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = 0.17, 95% CI 2-sided [0.01 to 0.32], Standard Error of Mean 0.08
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.51, 95% CI 2-sided [-0.66 to -0.35], Standard Error of Mean 0.08
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.56, 95% CI 2-sided [-0.72 to -0.41], Standard Error of Mean 0.08
Statistical Analysis 7: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.041, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.16, 95% CI 2-sided [-0.32 to -0.01], Standard Error of Mean 0.08
Statistical Analysis 8: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.006, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.22, 95% CI 2-sided [-0.38 to -0.06], Standard Error of Mean 0.08
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.44, 95% CI 2-sided [-0.60 to -0.27], Standard Error of Mean 0.08
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.45, 95% CI 2-sided [-0.62 to -0.29], Standard Error of Mean 0.08
Statistical Analysis 11: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p = 0.011, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.22, 95% CI 2-sided [-0.38 to -0.05], Standard Error of Mean 0.08
Statistical Analysis 12: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p = 0.006, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.23, 95% CI 2-sided [-0.40 to -0.07], Standard Error of Mean 0.08
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.43, 95% CI 2-sided [-0.60 to -0.26], Standard Error of Mean 0.08
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.31, 95% CI 2-sided [-0.48 to -0.14], Standard Error of Mean 0.08
Statistical Analysis 15: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.26, 95% CI 2-sided [-0.42 to -0.09], Standard Error of Mean 0.08
Statistical Analysis 16: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.105, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.14, 95% CI 2-sided [-0.30 to 0.03], Standard Error of Mean 0.08

9. Secondary Outcome: Change From Baseline in Patient Global Assessment of Osteoarthritis at Week 2, 4, 8 and 12: Last Observation Carried Forward (LOCF)
Description: as for outcome 3
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 198 | 201 | 202 | 200
units on a scale
  Baseline | 3.41 (0.61) | 3.41 (0.59) | 3.39 (0.55) | 3.44 (0.62)
  Change at Week 2 | -0.53 (0.78) | -0.69 (0.91) | -0.68 (0.90) | -0.89 (0.94)
  Change at Week 4 | -0.54 (0.76) | -1.01 (1.01) | -1.10 (0.91) | -0.91 (0.85)
  Change at Week 8 | -0.56 (0.83) | -0.96 (1.00) | -1.05 (0.95) | -0.81 (0.95)
  Change at Week 12 | -0.63 (0.83) | -1.01 (1.04) | -0.98 (0.96) | -0.82 (0.89)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.045, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.16, 95% CI 2-sided [-0.32 to -0.00], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.030, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.18, 95% CI 2-sided [-0.33 to -0.02], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.027, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = 0.18, 95% CI 2-sided [0.02 to 0.34], Standard Error of Mean 0.08
Statistical Analysis 4: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.040, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = 0.17, 95% CI 2-sided [0.01 to 0.32], Standard Error of Mean 0.08
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.48, 95% CI 2-sided [-0.64 to -0.32], Standard Error of Mean 0.08
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.58, 95% CI 2-sided [-0.74 to -0.42], Standard Error of Mean 0.08
Statistical Analysis 7: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.094, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.14, 95% CI 2-sided [-0.30 to 0.02], Standard Error of Mean 0.08
Statistical Analysis 8: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.24, 95% CI 2-sided [-0.40 to -0.08], Standard Error of Mean 0.08
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.40, 95% CI 2-sided [-0.57 to -0.23], Standard Error of Mean 0.08
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.51, 95% CI 2-sided [-0.68 to -0.35], Standard Error of Mean 0.08
Statistical Analysis 11: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p = 0.032, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.18, 95% CI 2-sided [-0.35 to -0.02], Standard Error of Mean 0.08
Statistical Analysis 12: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.29, 95% CI 2-sided [-0.46 to -0.13], Standard Error of Mean 0.08
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.38, 95% CI 2-sided [-0.54 to -0.21], Standard Error of Mean 0.08
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.36, 95% CI 2-sided [-0.52 to -0.19], Standard Error of Mean 0.08
Statistical Analysis 15: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.012, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.21, 95% CI 2-sided [-0.38 to -0.05], Standard Error of Mean 0.08
Statistical Analysis 16: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.021, ANCOVA — P-value was based on ANCOVA from pairwise comparisons; LS mean difference = -0.20, 95% CI 2-sided [-0.36 to -0.03], Standard Error of Mean 0.08

10. Secondary Outcome: Percentage of Responders For Outcome Measures in Rheumatology- Osteoarthritis Research Society International (OMERACT-OARSI): Baseline Observation Carried Forward (BOCF)
Description: A participant was considered as an OMERACT-OARSI responder: if the improvement from baseline to week of interest was greater than or equal to (>=) 50 percent and >=2 units in WOMAC pain or physical function subscale; if improvement from baseline to week of interest was >=20 percent and >=1 unit in at least 2 of the following: a) WOMAC pain subscale, b) WOMAC physical function subscale, c) PGA of osteoarthritis. WOMAC pain subscale assess amount of pain experienced (score: 0 [minimum pain] to 10 [maximum pain], higher score = more pain), WOMAC physical function subscale assess degree of difficulty experienced (score: 0 [minimum difficulty] to 10 [maximum difficulty], higher score = higher difficulty) and PGA of osteoarthritis (score: 1 [minimum affected] to 5 [maximum affected], higher score = worse condition). Percentage of participants who were OMERACT-OARSI responder were reported in this outcome measure.
Time Frame: Weeks 2, 4, 8, 12, 16
Population: mITT population included all participants who received at least 1 dose of the study drug, except those with concerns about data integrity at 1 of the study centers. BOCF method was used to impute missing values.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 200 | 202 | 203 | 200
percentage of participants
  Week 2 | 55.3 | 61.9 | 69.8 | 67.0
  Week 4 | 53.3 | 72.3 | 76.2 | 69.5
  Week 8 | 50.3 | 72.8 | 72.8 | 67.0
  Week 12 | 48.7 | 70.8 | 66.8 | 62.5
  Week 16 | 50.3 | 66.3 | 63.9 | 61.0

11. Secondary Outcome: Percentage of Responders For Outcome Measures in Rheumatology- Osteoarthritis Research Society International (OMERACT-OARSI): Last Observation Carried Forward (LOCF)
Description: as for outcome 10
Time Frame: Week 2, 4, 8, 12, 16
Population: mITT population included all participants who received at least 1 dose of the study drug, except those with concerns about data integrity at 1 of the study centers. LOCF method was used to impute missing values.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 200 | 202 | 203 | 200
percentage of participants
  Week 2 | 55.3 | 61.9 | 69.8 | 67.0
  Week 4 | 56.3 | 73.8 | 81.2 | 70.5
  Week 8 | 56.3 | 76.7 | 81.7 | 70.0
  Week 12 | 60.8 | 77.2 | 80.2 | 69.0
  Week 16 | 61.8 | 75.2 | 80.2 | 70.0

12. Secondary Outcome: Percentage of Participants With at Least 30 Percent, and 50 Percent Reduction in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms in participants with osteoarthritis of knee. WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in the index knee during past 48 hours. It is calculated as mean of the scores from 5 individual questions scored on a numerical rating scale of 0 (minimum pain) to 10 (maximum pain), where higher scores indicate more pain. An overall possible WOMAC pain subscale score range is of 0 (minimum pain) to 10 (maximum pain), where higher scores indicate more pain. Percentage of participants with at least 30 percent and 50 percent reduction in WOMAC pain subscale were reported in this outcome measure.
Time Frame: Week 2, 4, 8, 12, 16
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 199 | 202 | 202 | 200
percentage of participants
  Week 2: >=30 percent reduction | 46.7 | 52.0 | 58.4 | 60.5
  Week 2: >=50 percent reduction | 29.6 | 36.1 | 41.6 | 44.5
  Week 4: >=30 percent reduction | 47.2 | 65.8 | 72.8 | 62.5
  Week 4: >=50 percent reduction | 30.7 | 52.0 | 60.9 | 48.5
  Week 8: >=30 percent reduction | 44.7 | 68.3 | 70.3 | 62.5
  Week 8: >=50 percent reduction | 31.7 | 53.0 | 60.4 | 46.0
  Week 12: >=30 percent reduction | 44.2 | 69.3 | 65.8 | 58.0
  Week 12: >=50 percent reduction | 32.7 | 57.4 | 57.9 | 46.5
  Week 16: >=30 percent reduction | 42.7 | 65.8 | 59.4 | 55.5
  Week 16: >=50 percent reduction | 31.2 | 52.0 | 52.0 | 41.5

13. Secondary Outcome: Percentage of Participants With at Least 30 Percent, and 50 Percent Reduction in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale: Last Observation Carried Forward (LOCF)
Description: as for outcome 12
Time Frame: Week 2, 4, 8, 12, 16
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 199 | 202 | 202 | 200
percentage of participants
  Week 2: >=30 percent reduction | 46.7 | 52.0 | 58.4 | 60.5
  Week 2: >=50 percent reduction | 29.6 | 36.1 | 41.6 | 44.5
  Week 4: >=30 percent reduction | 51.3 | 66.8 | 76.7 | 63.5
  Week 4: >=50 percent reduction | 32.7 | 52.0 | 63.4 | 49.5
  Week 8: >=30 percent reduction | 51.8 | 71.3 | 78.2 | 65.0
  Week 8: >=50 percent reduction | 35.2 | 55.0 | 65.3 | 48.0
  Week 12: >=30 percent reduction | 56.8 | 73.8 | 77.2 | 64.5
  Week 12: >=50 percent reduction | 39.7 | 59.9 | 64.9 | 51.0
  Week 16: >=30 percent reduction | 54.3 | 73.3 | 73.3 | 65.5
  Week 16: >=50 percent reduction | 37.7 | 55.9 | 61.9 | 47.5

14. Secondary Outcome: Percentage of Participants With at Least 2 Points Improvement From Baseline in Patient Global Assessment (PGA) of Osteoarthritis: Baseline Observation Carried Forward (BOCF)
Description: Participants answered: "Considering all the ways the osteoarthritis in your index knee affects you, how are you doing today?" Participants responded on the scale ranging from 1 (minimum affected) to 5 (maximum affected), where 1= very good, 2= good, 3= fair, 4= poor and 5= very poor. Higher scores indicate worse condition. Percentage of participants with at least 2 points improvement from baseline in PGA of osteoarthritis at specified weeks were reported.
Time Frame: Baseline, Week 2, 4, 8, 12, 16
Population: mITT population included all participants who received at least 1 dose of the study drug, except those with concerns about data integrity at 1 of the study centers. BOCF method was used to impute missing values. Here, 'Number Analyzed' signifies number of participants evaluable at specific time points.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 200 | 202 | 203 | 200
percentage of participants
  Week 2: number analyzed (Participants) | 200 | 202 | 202 | 200
  Week 2 | 11.0 | 17.8 | 16.8 | 25.5
  Week 4 | 9.0 | 29.7 | 30.0 | 22.0
  Week 8 | 9.5 | 29.2 | 28.6 | 19.5
  Week 12: number analyzed (Participants) | 200 | 202 | 202 | 200
  Week 12 | 12.5 | 31.7 | 24.8 | 18.0
  Week 16: number analyzed (Participants) | 200 | 202 | 202 | 200
  Week 16 | 13.5 | 25.2 | 19.8 | 19.5

15. Secondary Outcome: Percentage of Participants With at Least 2 Points Improvement From Baseline in Patient Global Assessment (PGA) of Osteoarthritis: Last Observation Carried Forward (LOCF)
Description: as for outcome 14
Time Frame: Baseline, Week 2, 4, 8, 12, 16
Population: mITT population included all participants who received at least 1 dose of the study drug, except those with concerns about data integrity at 1 of the study centers. LOCF method was used to impute missing values. Here, 'Number Analyzed' signifies number of participants evaluable at specific time points.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 200 | 202 | 203 | 200
percentage of participants
  Week 2: number analyzed (Participants) | 200 | 202 | 202 | 200
  Week 2 | 11.0 | 17.8 | 16.8 | 25.5
  Week 4 | 9.0 | 29.7 | 31.5 | 22.5
  Week 8 | 10.0 | 29.7 | 31.5 | 20.0
  Week 12 | 14.5 | 33.7 | 29.1 | 20.5
  Week 16 | 16.0 | 27.7 | 24.6 | 22.5

16. Secondary Outcome: Percentage of Participants With Cumulative Reduction From Baseline up to Week 16 in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms in participants with osteoarthritis of knee. WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in the index knee during past 48 hours. It is calculated as mean of the scores from 5 individual questions scored on a numerical rating scale of 0 (minimum pain) to 10 (maximum pain), where higher scores indicate more pain. An overall possible WOMAC pain subscale score range is of 0 (minimum pain) to 10 (maximum pain), where higher scores indicate more pain. Percentage of participants with cumulative reduction (greater than 0 percent [%]; >= 10 %, 20 %, 30 %, 40 %, 50 %, 60 %, 70 %, 80 % and 90%; = 100 %) in WOMAC pain subscale from Baseline up to Week 16 were reported.
Time Frame: Baseline up to Week 16
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 199 | 202 | 202 | 200
percentage of participants
  Greater than (>) 0 percent | 57.3 | 73.3 | 69.3 | 71.5
  >=10 percent | 54.3 | 71.8 | 66.3 | 68.0
  >=20 percent | 50.8 | 68.3 | 64.4 | 62.0
  >=30 percent | 42.7 | 65.8 | 59.4 | 55.5
  >=40 percent | 36.7 | 60.4 | 56.4 | 50.0
  >=50 percent | 31.2 | 52.0 | 52.0 | 41.5
  >=60 percent | 27.6 | 49.5 | 47.0 | 35.5
  >=70 percent | 22.1 | 39.1 | 37.6 | 26.0
  >=80 percent | 14.6 | 29.2 | 25.2 | 18.0
  >=90 percent | 8.0 | 18.8 | 17.8 | 11.0
  100 percent | 3.0 | 8.4 | 7.4 | 4.0

17. Secondary Outcome: Percentage of Participants With Cumulative Reduction From Baseline up to Week 16 in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score: Last Observation Carried Forward (LOCF)
Description: as for outcome 16
Time Frame: Baseline up to Week 16
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 199 | 202 | 202 | 200
percentage of participants
  >0 percent | 82.4 | 87.6 | 92.1 | 91.5
  >=10 percent | 75.4 | 83.2 | 86.1 | 83.0
  >=20 percent | 66.8 | 77.7 | 82.2 | 73.0
  >=30 percent | 54.3 | 73.3 | 73.3 | 65.5
  >=40 percent | 45.7 | 66.3 | 68.3 | 57.0
  >=50 percent | 37.7 | 55.9 | 61.9 | 47.5
  >=60 percent | 31.7 | 53.0 | 54.5 | 41.0
  >=70 percent | 24.6 | 41.6 | 43.6 | 30.0
  >=80 percent | 15.6 | 29.7 | 28.7 | 21.5
  >=90 percent | 9.0 | 19.3 | 19.8 | 13.0
  100 percent | 3.5 | 8.9 | 7.9 | 5.0

18. Secondary Outcome: Change From Baseline for the Average Pain Score in the Index Knee at Week 2, 4, 8, 12 and 16: Baseline Observation Carried Forward (BOCF)
Description: Participants assessed daily average pain score in the index knee using a scale ranging from 0 (no pain) to 10 (maximum pain), where higher scores indicate more pain. A weekly mean was calculated using the daily average index knee pain scores within each specified study week.
Time Frame: Baseline, Week 2, 4, 8, 12, 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 197 | 200 | 199 | 199
units on a scale
  Baseline | 6.46 (1.83) | 6.51 (1.98) | 6.58 (1.70) | 6.70 (1.99)
  Change at Week 2 | -1.23 (2.08) | -1.80 (2.45) | -2.08 (2.20) | -2.39 (2.28)
  Change at Week 4 | -1.34 (2.27) | -2.46 (2.52) | -2.91 (2.52) | -2.33 (2.33)
  Change at Week 8 | -1.48 (2.34) | -2.52 (2.72) | -2.92 (2.61) | -2.42 (2.63)
  Change at Week 12 | -1.53 (2.32) | -2.82 (2.80) | -2.79 (2.63) | -2.30 (2.68)
  Change at Week 16 | -1.44 (2.25) | -2.54 (2.77) | -2.48 (2.67) | -2.21 (2.53)

19. Secondary Outcome: Change From Baseline for the Average Pain Score in the Index Knee at Week 2, 4, 8, 12 and 16: Last Observation Carried Forward (LOCF)
Description: as for outcome 18
Time Frame: Baseline, Week 2, 4, 8, 12, 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 200 | 202 | 203 | 200
units on a scale
  Baseline | 6.43 (1.84) | 6.51 (1.97) | 6.60 (1.70) | 6.69 (1.99)
  Change at Week 2: number analyzed (Participants) | 197 | 200 | 199 | 199
  Change at Week 2 | -1.25 (2.10) | -1.84 (2.46) | -2.09 (2.20) | -2.39 (2.28)
  Change at Week 4: number analyzed (Participants) | 197 | 200 | 199 | 199
  Change at Week 4 | -1.33 (2.38) | -2.58 (2.54) | -2.96 (2.54) | -2.40 (2.32)
  Change at Week 8: number analyzed (Participants) | 197 | 200 | 199 | 199
  Change at Week 8 | -1.45 (2.51) | -2.66 (2.69) | -3.13 (2.58) | -2.49 (2.62)
  Change at Week 12: number analyzed (Participants) | 197 | 200 | 199 | 199
  Change at Week 12 | -1.68 (2.70) | -3.03 (2.73) | -3.20 (2.59) | -2.67 (2.67)
  Change at Week 16: number analyzed (Participants) | 197 | 200 | 199 | 199
  Change at Week 16 | -1.67 (2.68) | -2.79 (2.75) | -2.96 (2.66) | -2.60 (2.56)

20. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale at Week 2, 4, 8, 12 and 16: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms in participants with osteoarthritis of knee. WOMAC stiffness subscale is a 2-item questionnaire used to assess the amount of stiffness experienced due to osteoarthritis in knee joint during past 48 hours. It is calculated as mean of the scores from 2 individual questions each scored on numerical rating scale of 0 (minimum stiffness) to 10 (maximum stiffness), where higher scores indicate greater stiffness. An overall possible WOMAC stiffness subscale score range is of 0 (minimum stiffness) to 10 (maximum stiffness), where higher scores indicate higher stiffness. Stiffness is defined as a sensation of decreased ease in moving the index knee.
Time Frame: Baseline, Week 2, 4, 8, 12, 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 199 | 202 | 202 | 200
units on a scale
  Baseline | 7.04 (1.88) | 7.17 (1.72) | 7.04 (1.75) | 7.02 (1.76)
  Change at Week 2 | -1.69 (2.36) | -2.63 (2.78) | -2.98 (2.63) | -2.81 (2.67)
  Change at Week 4 | -1.76 (2.44) | -3.40 (2.81) | -3.84 (2.73) | -2.87 (2.63)
  Change at Week 8 | -1.77 (2.26) | -3.42 (2.73) | -3.68 (2.81) | -2.60 (2.76)
  Change at Week 12 | -1.82 (2.40) | -3.73 (2.88) | -3.46 (2.94) | -2.62 (2.70)
  Change at Week 16 | -1.72 (2.27) | -3.33 (2.84) | -3.16 (2.93) | -2.31 (2.68)

21. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale at Week 2, 4, 8, 12 and 16: Last Observation Carried Forward (LOCF)
Description: as for outcome 20
Time Frame: Baseline, Week 2, 4, 8, 12, 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 199 | 202 | 202 | 200
units on a scale
  Baseline | 7.04 (1.88) | 7.17 (1.72) | 7.04 (1.75) | 7.02 (1.76)
  Change at Week 2 | -1.69 (2.36) | -2.63 (2.78) | -2.98 (2.63) | -2.81 (2.67)
  Change at Week 4 | -1.81 (2.53) | -3.42 (2.89) | -3.95 (2.63) | -2.92 (2.62)
  Change at Week 8 | -1.95 (2.34) | -3.57 (2.78) | -4.00 (2.68) | -2.72 (2.78)
  Change at Week 12 | -2.18 (2.54) | -3.99 (2.86) | -4.05 (2.70) | -2.91 (2.75)
  Change at Week 16 | -2.07 (2.43) | -3.73 (2.80) | -3.91 (2.68) | -2.73 (2.75)

22. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Average Score at Week 2, 4, 8, 12 and 16: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms in participants with osteoarthritis of knee. WOMAC pain subscale assess amount of pain experienced (score: 0 [minimum pain] to 10 [maximum pain], higher score = more pain), WOMAC physical function subscale assess degree of difficulty experienced (score: 0 [minimum difficulty] to 10 [maximum difficulty], higher score = higher difficulty) and WOMAC stiffness subscale assess the amount of stiffness experienced (score: 0 [minimum stiffness] to 10 [maximum stiffness], higher score = higher stiffness). WOMAC average score is the mean of WOMAC pain, physical function and stiffness subscale scores, giving an overall possible WOMAC average score range of 0 (minimum difficulty) to 10 (maximum difficulty), where higher scores indicate worse response.
Time Frame: Baseline, Week 2, 4, 8, 12, 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 199 | 202 | 202 | 200
units on a scale
  Baseline | 7.03 (1.48) | 7.11 (1.46) | 7.05 (1.38) | 7.02 (1.37)
  Change at Week 2 | -1.99 (2.12) | -2.56 (2.47) | -2.91 (2.34) | -2.86 (2.35)
  Change at Week 4 | -2.02 (2.21) | -3.35 (2.49) | -3.82 (2.49) | -3.02 (2.33)
  Change at Week 8 | -2.03 (2.14) | -3.41 (2.49) | -3.70 (2.60) | -2.81 (2.49)
  Change at Week 12 | -2.00 (2.35) | -3.69 (2.69) | -3.48 (2.77) | -2.75 (2.51)
  Change at Week 16 | -1.95 (2.30) | -3.35 (2.66) | -3.12 (2.69) | -2.52 (2.43)

23. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Average Score at Week 2, 4, 8, 12 and 16: Last Observation Carried Forward (LOCF)
Description: as for outcome 22
Time Frame: Baseline, Week 2, 4, 8, 12, 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 199 | 202 | 202 | 200
units on a scale
  Baseline | 7.03 (1.48) | 7.11 (1.46) | 7.05 (1.38) | 7.02 (1.37)
  Change at Week 2 | -1.99 (2.12) | -2.56 (2.47) | -2.91 (2.34) | -2.86 (2.35)
  Change at Week 4 | -2.13 (2.23) | -3.36 (2.54) | -3.94 (2.38) | -3.06 (2.31)
  Change at Week 8 | -2.23 (2.18) | -3.52 (2.49) | -4.00 (2.41) | -2.94 (2.45)
  Change at Week 12 | -2.44 (2.36) | -3.89 (2.61) | -4.02 (2.46) | -3.06 (2.47)
  Change at Week 16 | -2.37 (2.33) | -3.67 (2.53) | -3.82 (2.38) | -2.96 (2.39)

24. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score When Walking on a Flat Surface at Week 2, 4, 8, 12 and 16: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms in participants with osteoarthritis of knee. Participants responded by using a numerical rating scale of 0 (no pain) to 10 (maximum pain) about the amount of pain they experienced when walking on a flat surface, where 0= no pain and 10= extreme pain. Higher score indicates more pain.
Time Frame: Baseline, Week 2, 4, 8, 12, 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 199 | 202 | 202 | 200
units on a scale
  Baseline | 7.22 (1.65) | 7.16 (1.79) | 7.08 (1.70) | 7.04 (1.71)
  Change at Week 2 | -2.40 (2.43) | -2.52 (2.72) | -2.96 (2.65) | -3.05 (2.60)
  Change at Week 4 | -2.36 (2.49) | -3.49 (2.67) | -3.89 (2.70) | -3.30 (2.48)
  Change at Week 8 | -2.41 (2.52) | -3.52 (2.78) | -3.80 (2.84) | -3.05 (2.72)
  Change at Week 12 | -2.28 (2.67) | -3.73 (2.91) | -3.50 (2.98) | -2.98 (2.77)
  Change at Week 16 | -2.26 (2.70) | -3.39 (3.00) | -3.10 (2.83) | -2.72 (2.63)

25. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score When Walking on a Flat Surface at Week 2, 4, 8, 12 and 16: Last Observation Carried Forward (LOCF)
Description: as for outcome 24
Time Frame: Baseline, Week 2, 4, 8, 12, 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 199 | 202 | 202 | 200
units on a scale
  Baseline | 7.22 (1.65) | 7.16 (1.79) | 7.08 (1.70) | 7.04 (1.71)
  Change at Week 2 | -2.40 (2.43) | -2.52 (2.72) | -2.96 (2.65) | -3.05 (2.60)
  Change at Week 4 | -2.58 (2.51) | -3.53 (2.65) | -4.02 (2.63) | -3.35 (2.44)
  Change at Week 8 | -2.71 (2.53) | -3.65 (2.74) | -4.11 (2.66) | -3.23 (2.65)
  Change at Week 12 | -2.87 (2.64) | -3.94 (2.78) | -4.01 (2.72) | -3.40 (2.66)
  Change at Week 16 | -2.84 (2.68) | -3.71 (2.83) | -3.77 (2.63) | -3.28 (2.50)

26. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score When Going Up or Down Stairs at Week 2, 4, 8, 12 and 16: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms in participants with osteoarthritis of knee. Participants responded by using a numerical rating scale of 0 (no pain) to 10 (maximum pain) about the amount of pain they experienced when going up or down stairs, where 0= no pain and 10= extreme pain. Higher score indicates more pain.
Time Frame: Baseline, Week 2, 4, 8, 12, 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 199 | 202 | 202 | 200
units on a scale
  Baseline | 8.24 (1.33) | 8.29 (1.43) | 8.15 (1.47) | 8.30 (1.35)
  Change at Week 2 | -2.19 (2.50) | -2.86 (2.78) | -3.10 (2.68) | -3.24 (2.75)
  Change at Week 4 | -2.18 (2.49) | -3.61 (2.72) | -4.18 (2.90) | -3.39 (2.76)
  Change at Week 8 | -2.15 (2.55) | -3.65 (2.89) | -3.98 (3.00) | -3.25 (2.86)
  Change at Week 12 | -2.14 (2.70) | -4.01 (3.00) | -3.79 (3.17) | -3.06 (2.96)
  Change at Week 16 | -2.21 (2.73) | -3.61 (3.05) | -3.38 (3.09) | -2.93 (2.77)

27. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score When Going Up or Down Stairs at Week 2, 4, 8, 12 and 16: Last Observation Carried Forward (LOCF)
Description: as for outcome 26
Time Frame: Baseline, Week 2, 4, 8, 12, 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 199 | 202 | 202 | 200
units on a scale
  Baseline | 8.24 (1.33) | 8.29 (1.43) | 8.15 (1.47) | 8.30 (1.35)
  Change at Week 2 | -2.19 (2.50) | -2.86 (2.78) | -3.10 (2.68) | -3.24 (2.75)
  Change at Week 4 | -2.30 (2.52) | -3.65 (2.70) | -4.33 (2.77) | -3.44 (2.73)
  Change at Week 8 | -2.38 (2.57) | -3.81 (2.82) | -4.36 (2.77) | -3.40 (2.84)
  Change at Week 12 | -2.61 (2.68) | -4.25 (2.83) | -4.35 (2.84) | -3.46 (2.91)
  Change at Week 16 | -2.65 (2.71) | -3.99 (2.84) | -4.10 (2.78) | -3.48 (2.69)

28. Secondary Outcome: Change From Baseline in Short-Form 36 Health Survey (SF-36) 8 Health Domains, Mental Component Aggregate and Physical Component Aggregate Scores at Week 12 and 16: Baseline Observation Carried Forward (BOCF)
Description: SF-36 health survey is a self-administered questionnaire that measures each of the following 8 health domains: domain 1= general health, domain 2= physical function, domain 3= role physical, domain 4= bodily pain, domain 5= vitality, domain 6= social function, domain 7= role emotional and domain 8= mental health. Total score for each of the 8 domains are scaled from 0 (minimum level of functioning) to 100 (maximum level of functioning). These 8 domains are also summarized as 2 summary scores: mental component aggregate (MCA) and physical component aggregate (PCA). Total score range for each of the 2 summary scores =0 (minimum level of functioning) to 100 (maximum level of functioning). Higher (8 domains and 2 summary) scores indicate a better health related quality of life.
Time Frame: Baseline, Week 12, 16
Population: mITT population included all participants who received at least 1 dose of the study drug, except those with concerns about data integrity at 1 of the study centers. BOCF method was used to impute missing values. Here, 'Number Analyzed' signifies number of participants evaluable for specific time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 200 | 202 | 203 | 200
units on a scale
  Baseline: Domain 1: number analyzed (Participants) | 199 | 201 | 201 | 200
  Baseline: Domain 1 | 66.03 (19.88) | 67.19 (17.71) | 67.64 (19.71) | 65.16 (19.77)
  Change at Week 12:Domain 1: number analyzed (Participants) | 199 | 201 | 201 | 200
  Change at Week 12:Domain 1 | 4.13 (11.47) | 6.33 (13.62) | 3.23 (11.60) | 4.12 (13.11)
  Change at Week 16:Domain 1: number analyzed (Participants) | 199 | 201 | 201 | 200
  Change at Week 16:Domain 1 | 3.42 (11.57) | 4.03 (14.02) | 3.31 (11.32) | 3.62 (12.40)
  Baseline: Domain 2: number analyzed (Participants) | 199 | 201 | 202 | 200
  Baseline: Domain 2 | 30.45 (19.83) | 32.69 (19.88) | 34.53 (18.96) | 31.93 (18.48)
  Change at Week 12:Domain 2: number analyzed (Participants) | 199 | 201 | 202 | 200
  Change at Week 12:Domain 2 | 10.15 (18.50) | 18.45 (22.97) | 17.47 (23.51) | 12.69 (19.68)
  Change at Week 16:Domain 2: number analyzed (Participants) | 199 | 201 | 201 | 200
  Change at Week 16:Domain 2 | 8.74 (17.38) | 15.38 (21.77) | 13.94 (22.15) | 11.08 (19.04)
  Baseline: Domain 3: number analyzed (Participants) | 199 | 201 | 202 | 200
  Baseline: Domain 3 | 43.62 (25.48) | 44.21 (26.10) | 46.50 (23.89) | 45.44 (25.54)
  Change at Week 12:Domain 3: number analyzed (Participants) | 199 | 201 | 202 | 200
  Change at Week 12:Domain 3 | 10.77 (22.74) | 20.00 (26.45) | 17.57 (25.61) | 13.03 (24.97)
  Change at Week 16:Domain 3: number analyzed (Participants) | 199 | 201 | 202 | 200
  Change at Week 16:Domain 3 | 9.64 (21.87) | 17.33 (27.01) | 15.10 (23.84) | 11.69 (22.79)
  Baseline: Domain 4: number analyzed (Participants) | 199 | 201 | 202 | 200
  Baseline: Domain 4 | 33.72 (17.09) | 33.65 (16.04) | 33.72 (14.85) | 34.02 (16.74)
  Change at Week 12:Domain 4: number analyzed (Participants) | 199 | 201 | 202 | 200
  Change at Week 12:Domain 4 | 13.67 (20.32) | 23.08 (23.15) | 21.07 (23.88) | 14.93 (20.47)
  Change at Week 16:Domain 4: number analyzed (Participants) | 199 | 201 | 202 | 200
  Change at Week 16:Domain 4 | 11.23 (18.48) | 18.99 (22.90) | 16.76 (21.85) | 13.19 (21.19)
  Baseline: Domain 5: number analyzed (Participants) | 198 | 201 | 202 | 200
  Baseline: Domain 5 | 53.09 (20.63) | 51.00 (21.81) | 52.32 (18.93) | 51.84 (20.54)
  Change at Week 12:Domain 5: number analyzed (Participants) | 198 | 201 | 202 | 200
  Change at Week 12:Domain 5 | 4.39 (12.54) | 10.29 (18.21) | 6.96 (16.19) | 7.19 (14.89)
  Change at Week 16:Domain 5: number analyzed (Participants) | 198 | 201 | 202 | 200
  Change at Week 16:Domain 5 | 3.98 (13.51) | 8.83 (17.22) | 7.52 (14.84) | 5.66 (14.86)
  Baseline: Domain 6: number analyzed (Participants) | 199 | 201 | 202 | 200
  Baseline: Domain 6 | 69.28 (27.86) | 68.53 (26.43) | 69.86 (25.08) | 67.94 (25.48)
  Change at Week 12:Domain 6: number analyzed (Participants) | 199 | 201 | 202 | 200
  Change at Week 12:Domain 6 | 9.05 (21.02) | 11.82 (25.32) | 8.48 (21.71) | 9.44 (20.84)
  Change at Week 16:Domain 6: number analyzed (Participants) | 199 | 201 | 202 | 200
  Change at Week 16:Domain 6 | 6.97 (20.78) | 11.63 (24.76) | 7.43 (18.80) | 8.00 (22.90)
  Baseline: Domain 7: number analyzed (Participants) | 199 | 201 | 202 | 200
  Baseline: Domain 7 | 70.69 (32.12) | 71.52 (29.63) | 72.94 (27.16) | 71.54 (29.22)
  Change at Week 12:Domain 7: number analyzed (Participants) | 199 | 201 | 201 | 200
  Change at Week 12:Domain 7 | 6.03 (19.98) | 9.00 (26.96) | 6.06 (18.70) | 4.88 (24.57)
  Change at Week 16:Domain 7: number analyzed (Participants) | 199 | 201 | 202 | 200
  Change at Week 16:Domain 7 | 4.61 (23.50) | 8.46 (23.88) | 4.21 (18.78) | 4.62 (21.99)
  Baseline: Domain 8: number analyzed (Participants) | 199 | 201 | 202 | 200
  Baseline: Domain 8 | 76.06 (18.01) | 75.80 (17.76) | 74.48 (17.95) | 74.91 (17.79)
  Change at Week 12:Domain 8: number analyzed (Participants) | 199 | 201 | 202 | 200
  Change at Week 12:Domain 8 | 2.94 (11.39) | 3.46 (16.38) | 3.66 (12.94) | 2.56 (13.50)
  Change at Week 16:Domain 8: number analyzed (Participants) | 199 | 201 | 202 | 200
  Change at Week 16:Domain 8 | 1.66 (13.81) | 3.21 (15.31) | 2.97 (12.37) | 2.31 (13.32)
  Baseline: MCA: number analyzed (Participants) | 198 | 201 | 201 | 200
  Baseline: MCA | 0.31 (1.27) | 0.26 (1.21) | 0.25 (1.15) | 0.24 (1.21)
  Change at Week 12: MCA: number analyzed (Participants) | 198 | 201 | 201 | 200
  Change at Week 12: MCA | 0.15 (0.70) | 0.16 (1.03) | 0.07 (0.76) | 0.11 (0.84)
  Change at Week 16: MCA: number analyzed (Participants) | 198 | 201 | 201 | 200
  Change at Week 16: MCA | 0.09 (0.81) | 0.19 (0.93) | 0.06 (0.71) | 0.10 (0.86)
  Baseline: PCA: number analyzed (Participants) | 198 | 201 | 201 | 200
  Baseline: PCA | -1.92 (0.74) | -1.85 (0.76) | -1.78 (0.72) | -1.86 (0.78)
  Change at Week 12: PCA: number analyzed (Participants) | 198 | 201 | 201 | 200
  Change at Week 12: PCA | 0.47 (0.74) | 0.88 (0.90) | 0.77 (0.93) | 0.59 (0.80)
  Change at Week 16: PCA: number analyzed (Participants) | 198 | 201 | 201 | 200
  Change at Week 16: PCA | 0.42 (0.73) | 0.71 (0.89) | 0.66 (0.87) | 0.51 (0.81)

29. Secondary Outcome: Change From Baseline in Short-Form 36 Health Survey (SF-36) 8 Health Domains, Mental Component Aggregate and Physical Component Aggregate Scores at Week 12 and 16: Last Observation Carried Forward (LOCF)
Description: as for outcome 28
Time Frame: Baseline, Week 12, 16
Population: mITT population included all participants who received at least 1 dose of the study drug, except those with concerns about data integrity at 1 of the study centers. LOCF method was used to impute missing values. Here, 'Number Analyzed' signifies number of participants evaluable for specific time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 200 | 202 | 203 | 200
units on a scale
  Baseline: Domain 1: number analyzed (Participants) | 199 | 201 | 201 | 200
  Baseline: Domain 1 | 66.03 (19.88) | 67.19 (17.71) | 67.64 (19.71) | 65.16 (19.77)
  Change at Week 12:Domain 1: number analyzed (Participants) | 199 | 201 | 201 | 200
  Change at Week 12:Domain 1 | 4.13 (11.47) | 6.33 (13.62) | 3.23 (11.60) | 4.12 (13.11)
  Change at Week 16:Domain 1: number analyzed (Participants) | 199 | 201 | 201 | 200
  Change at Week 16:Domain 1 | 3.61 (11.72) | 4.76 (14.31) | 3.47 (11.73) | 4.23 (13.16)
  Baseline: Domain 2: number analyzed (Participants) | 199 | 201 | 202 | 200
  Baseline: Domain 2 | 30.45 (19.83) | 32.69 (19.88) | 34.53 (18.96) | 31.93 (18.48)
  Change at Week 12:Domain 2: number analyzed (Participants) | 199 | 201 | 202 | 200
  Change at Week 12:Domain 2 | 10.15 (18.50) | 18.45 (22.97) | 17.47 (23.51) | 12.69 (19.68)
  Change at Week 16:Domain 2: number analyzed (Participants) | 199 | 201 | 202 | 200
  Change at Week 16:Domain 2 | 9.80 (18.40) | 17.14 (21.58) | 15.48 (22.71) | 11.80 (19.21)
  Baseline: Domain 3: number analyzed (Participants) | 199 | 201 | 202 | 200
  Baseline: Domain 3 | 43.62 (25.48) | 44.21 (26.10) | 46.50 (23.89) | 45.44 (25.54)
  Change at Week 12:Domain 3: number analyzed (Participants) | 199 | 201 | 202 | 200
  Change at Week 12:Domain 3 | 10.77 (22.74) | 20.00 (26.45) | 17.57 (25.61) | 13.03 (24.97)
  Change at Week 16:Domain 3: number analyzed (Participants) | 199 | 201 | 202 | 200
  Change at Week 16:Domain 3 | 10.05 (22.09) | 19.04 (26.83) | 17.23 (24.53) | 12.59 (23.53)
  Baseline: Domain 4: number analyzed (Participants) | 199 | 201 | 202 | 200
  Baseline: Domain 4 | 33.72 (17.09) | 33.65 (16.04) | 33.72 (14.85) | 34.02 (16.74)
  Change at Week 12:Domain 4: number analyzed (Participants) | 199 | 201 | 202 | 200
  Change at Week 12:Domain 4 | 13.67 (20.32) | 23.08 (23.15) | 21.07 (23.88) | 14.93 (20.47)
  Change at Week 16:Domain 4: number analyzed (Participants) | 199 | 201 | 202 | 200
  Change at Week 16:Domain 4 | 11.53 (18.48) | 21.16 (22.93) | 19.19 (22.71) | 14.50 (21.46)
  Baseline: Domain 5: number analyzed (Participants) | 198 | 201 | 202 | 200
  Baseline: Domain 5 | 53.09 (20.63) | 51.00 (21.81) | 52.32 (18.93) | 51.84 (20.54)
  Change at Week 12:Domain 5: number analyzed (Participants) | 198 | 201 | 202 | 200
  Change at Week 12:Domain 5 | 4.39 (12.54) | 10.29 (18.21) | 6.96 (16.19) | 7.19 (14.89)
  Change at Week 16:Domain 5: number analyzed (Participants) | 198 | 201 | 202 | 200
  Change at Week 16:Domain 5 | 4.36 (14.22) | 9.20 (17.50) | 8.35 (15.53) | 6.22 (15.43)
  Baseline: Domain 6: number analyzed (Participants) | 199 | 201 | 202 | 200
  Baseline: Domain 6 | 69.28 (27.86) | 68.53 (26.43) | 69.86 (25.08) | 67.94 (25.48)
  Change at Week 12:Domain 6: number analyzed (Participants) | 199 | 201 | 202 | 200
  Change at Week 12:Domain 6 | 9.05 (21.02) | 11.82 (25.32) | 8.48 (21.71) | 9.44 (20.84)
  Change at Week 16:Domain 6: number analyzed (Participants) | 199 | 201 | 202 | 200
  Change at Week 16:Domain 6 | 7.29 (20.84) | 12.13 (25.06) | 8.79 (20.15) | 8.81 (23.57)
  Baseline: Domain 7: number analyzed (Participants) | 199 | 201 | 202 | 200
  Baseline: Domain 7 | 70.69 (32.12) | 71.52 (29.63) | 72.94 (27.16) | 71.54 (29.22)
  Change at Week 12:Domain 7: number analyzed (Participants) | 199 | 201 | 202 | 200
  Change at Week 12:Domain 7 | 6.03 (19.98) | 9.00 (26.96) | 6.06 (18.70) | 4.88 (24.57)
  Change at Week 16:Domain 7: number analyzed (Participants) | 199 | 201 | 202 | 200
  Change at Week 16:Domain 7 | 4.90 (23.69) | 8.91 (24.12) | 5.57 (20.13) | 4.92 (23.06)
  Baseline: Domain 8: number analyzed (Participants) | 199 | 201 | 202 | 200
  Baseline: Domain 8 | 76.06 (18.01) | 75.80 (17.76) | 74.48 (17.95) | 74.91 (17.79)
  Change at Week 12:Domain 8: number analyzed (Participants) | 199 | 201 | 202 | 200
  Change at Week 12:Domain 8 | 2.94 (11.39) | 3.46 (16.38) | 3.66 (12.94) | 2.56 (13.50)
  Change at Week 16:Domain 8: number analyzed (Participants) | 199 | 201 | 202 | 200
  Change at Week 16:Domain 8 | 1.93 (14.36) | 3.21 (15.72) | 3.56 (13.42) | 2.59 (13.78)
  Baseline: MCA: number analyzed (Participants) | 193 | 201 | 201 | 200
  Baseline: MCA | 0.31 (1.27) | 0.26 (1.21) | 0.25 (1.15) | 0.24 (1.21)
  Change at Week 12: MCA: number analyzed (Participants) | 198 | 201 | 201 | 200
  Change at Week 12: MCA | 0.15 (0.70) | 0.16 (1.03) | 0.07 (0.76) | 0.11 (0.84)
  Change at Week 16: MCA: number analyzed (Participants) | 198 | 201 | 201 | 200
  Change at Week 16: MCA | 0.10 (0.83) | 0.17 (0.95) | 0.10 (0.76) | 0.11 (0.90)
  Baseline: PCA: number analyzed (Participants) | 198 | 201 | 201 | 200
  Baseline: PCA | -1.92 (0.74) | -1.85 (0.76) | -1.78 (0.72) | -1.86 (0.78)
  Change at Week 12: PCA: number analyzed (Participants) | 198 | 201 | 201 | 200
  Change at Week 12: PCA | 0.47 (0.74) | 0.88 (0.90) | 0.77 (0.93) | 0.59 (0.80)
  Change at Week 16: PCA: number analyzed (Participants) | 198 | 201 | 201 | 200
  Change at Week 16: PCA | 0.45 (0.74) | 0.80 (0.88) | 0.73 (0.88) | 0.56 (0.82)

30. Secondary Outcome: Time to Discontinuation Due to Lack of Efficacy
Description: Median time to discontinuation due to lack of efficacy was estimated using Kaplan-Meier method.
Time Frame: Baseline up to Week 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of the study drug.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 208 | 206 | 208 | 206
days | NA [NA to NA] — Median and full range cannot be estimated due to less number of participants with events. | NA [NA to NA] — Median and full range cannot be estimated due to less number of participants with events. | NA [NA to NA] — Median and full range cannot be estimated due to less number of participants with events. | NA [NA to NA] — Median and full range cannot be estimated due to less number of participants with events.

31. Secondary Outcome: Percentage of Participants Who Used Rescue Medication
Description: In case of inadequate pain relief for osteoarthritis, acetaminophen up to 4000 mg per day up to 3 days in a week could be taken as rescue medication. Percentage of participants with any use of rescue medication during the specified study week were summarized.
Time Frame: Week 2, 4, 8, 12, 16
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 200 | 202 | 203 | 200
percentage of participants
  Week 2 | 62.5 | 47.3 | 58.6 | 49.7
  Week 4 | 59.5 | 35.3 | 38.9 | 47.0
  Week 8 | 53.5 | 35.8 | 33.0 | 40.0
  Week 12 | 42.5 | 29.4 | 30.5 | 32.0
  Week 16 | 40.5 | 26.9 | 25.1 | 36.0

32. Secondary Outcome: Number of Days Participants Used Rescue Medication
Description: In case of inadequate pain relief for osteoarthritis, acetaminophen up to 4000 mg per day up to 3 days in a week could be taken as rescue medication. Number of days participants used any of the rescue medication, during the specified week were summarized.
Time Frame: Week 2, 4, 8, 12, 16
Population: as for outcome 15
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 200 | 202 | 203 | 200
days
  Week 2: number analyzed (Participants) | 200 | 201 | 203 | 199
  Week 2 | 1 [0 to 7] | 0 [0 to 7] | 1 [0 to 7] | 0 [0 to 7]
  Week 4: number analyzed (Participants) | 200 | 201 | 203 | 200
  Week 4 | 1 [0 to 7] | 0 [0 to 7] | 0 [0 to 7] | 0 [0 to 7]
  Week 8: number analyzed (Participants) | 200 | 201 | 203 | 200
  Week 8 | 1 [0 to 7] | 0 [0 to 7] | 0 [0 to 7] | 0 [0 to 7]
  Week 12: number analyzed (Participants) | 200 | 201 | 203 | 200
  Week 12 | 0 [0 to 7] | 0 [0 to 7] | 0 [0 to 7] | 0 [0 to 7]
  Week 16: number analyzed (Participants) | 200 | 201 | 203 | 200
  Week 16 | 0 [0 to 7] | 0 [0 to 7] | 0 [0 to 7] | 0 [0 to 7]

33. Secondary Outcome: Amount of Rescue Medication Taken
Description: In case of inadequate pain relief for osteoarthritis, acetaminophen up to 4000 mg per day up to 3 days in a week could be taken as rescue medication. The total dosage of acetaminophen in mg used during the specified week were summarized.
Time Frame: Week 2, 4, 8, 12, 16
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 200 | 202 | 203 | 200
mg
  Week 2: number analyzed (Participants) | 200 | 201 | 203 | 199
  Week 2 | 3512.50 (5086.79) | 2644.28 (4867.40) | 2546.80 (3691.91) | 2025.13 (3468.75)
  Week 4: number analyzed (Participants) | 200 | 201 | 203 | 200
  Week 4 | 3492.50 (5755.81) | 1773.63 (3849.64) | 1795.57 (4134.95) | 2210.00 (3887.99)
  Week 8: number analyzed (Participants) | 200 | 201 | 203 | 200
  Week 8 | 3320.00 (5384.01) | 1684.08 (3506.56) | 1423.65 (3833.84) | 1987.50 (3967.02)
  Week 12: number analyzed (Participants) | 200 | 201 | 203 | 200
  Week 12 | 2857.50 (5617.94) | 1238.81 (3024.10) | 1504.93 (4054.39) | 1800.00 (4034.40)
  Week 16: number analyzed (Participants) | 200 | 201 | 203 | 200
  Week 16 | 2860.00 (5948.73) | 1427.86 (3733.77) | 1458.13 (4081.41) | 1872.50 (3967.52)

34. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) And Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Week 24 that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Day 1 (Baseline) up to Week 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 208 | 206 | 208 | 206
Participants
  Adverse Events | 99 | 107 | 122 | 104
  Serious Adverse Events | 8 | 7 | 6 | 5

35. Other Pre Specified Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Hemoglobin(Hgb),hematocrit,red blood cell(RBC):less than(<)0.8*lower limit of normal(LLN),MCV,MCH,MCHC<0.9*LLN or >1.1*ULN,platelet:<0.5*LLN or >1.75*upper limit of normal(ULN),white blood cell(WBC):<0.6*LLN or >1.5*ULN,lymphocyte,neutrophil,total neutrophil:<0.8*LLN or>1.2*ULN,basophil,eosinophil,monocyte:>1.2*ULN;total,direct bilirubin>1.5*ULN,aspartate aminotransferase,alanine aminotransferase,gamma-glutamyl transferase,LDH,alkaline phosphatase:> 3.0*ULN,total protein,albumin:<0.8*LLN or >1.2*ULN;blood urea nitrogen,creatinine:>1.3*ULN,uric acid>1.2*ULN;cholesterol,triglycerides>1.3*ULN;sodium <0.95*LLN or >1.05*ULN,potassium,chloride,calcium,magnesium,bicarbonate:<0.9*LLN or >1.1*ULN,phosphate<0.8*LLN or>1.2*ULN;glucose <0.6*LLN or >1.5*ULN,glycosylated Hgb >1.3*ULN,creatine kinase>2.0*ULN;urine(specific gravity <1.003or>1.030,pH <4.5or>8,glucose,ketone,protein,blood/Hgb,bilirubin,leukocyte esterase,crystals>=1,RBC,WBC >1.5*ULN,epithelial cell>=6,casts,hyaline cast>1,bacteria>20).
Time Frame: Day 1 (Baseline) up to Week 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of the study drug. Here, 'N' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 203 | 203 | 202 | 205
Participants | 146 | 155 | 139 | 162

36. Other Pre Specified Outcome: Number of Participants With 12-Lead Electrocardiogram (ECG) Abnormalities
Description: Criteria for potential clinical concern in ECG parameters are: Criterion 1= maximum QTcB interval (Bazett's correction) in range of 450 millisecond (msec) to less than 480 msec, Criterion 2= maximum QTcB interval in range of 480 msec to less than 500 msec, Criterion 3= maximum QTcB interval >= 500 msec; Criterion 4= maximum QTcF interval (Fridericia's correction) in range of 450 msec to less than 480 msec, Criterion 5= maximum QTcF interval in range of 480 msec to less than 500 msec, Criterion 6= maximum QTcF interval >= 500 msec, Criterion 7= maximum QTcB interval increase from baseline in range of 30 msec to less than 60 msec, Criterion 8= maximum QTcB interval increase >=60 msec, Criterion 9= maximum QTcF interval increase from baseline in range of 30 msec to less than 60 msec, Criterion 10= maximum QTcF interval increase >=60 msec.
Time Frame: Day 1 (Baseline) up to Week 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of the study drug. Here, 'Number Analyzed' signifies number of participants evaluable for specific time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 208 | 206 | 208 | 206
Participants
  Criterion 1: number analyzed (Participants) | 208 | 206 | 207 | 204
  Criterion 1 | 35 | 39 | 38 | 45
  Criterion 2: number analyzed (Participants) | 208 | 206 | 207 | 204
  Criterion 2 | 8 | 3 | 5 | 1
  Criterion 3: number analyzed (Participants) | 208 | 206 | 207 | 204
  Criterion 3 | 1 | 0 | 3 | 1
  Criterion 4: number analyzed (Participants) | 208 | 206 | 207 | 204
  Criterion 4 | 13 | 16 | 13 | 9
  Criterion 5: number analyzed (Participants) | 208 | 206 | 207 | 204
  Criterion 5 | 1 | 3 | 2 | 2
  Criterion 6: number analyzed (Participants) | 208 | 206 | 207 | 204
  Criterion 6 | 1 | 0 | 2 | 0
  Criterion 7: number analyzed (Participants) | 205 | 203 | 203 | 203
  Criterion 7 | 29 | 25 | 28 | 27
  Criterion 8: number analyzed (Participants) | 205 | 203 | 203 | 203
  Criterion 8 | 2 | 2 | 3 | 1
  Criterion 9: number analyzed (Participants) | 205 | 203 | 203 | 203
  Criterion 9 | 13 | 18 | 21 | 21
  Criterion 10: number analyzed (Participants) | 205 | 203 | 203 | 203
  Criterion 10 | 2 | 1 | 1 | 1

37. Other Pre Specified Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 2, 4, 8, 12, 16 and 24
Description: NIS is a standardized instrument used to evaluate participant for signs of peripheral neuropathy. NIS is the sum of scores of 37 items from both the left and right side, where 24 items scored from 0 (normal function) to 4 (extreme abnormal function), higher score indicates higher abnormality and 13 items scored from 0 (normal function) to 2 (extreme abnormal function), higher score indicates higher abnormality. NIS possible overall score ranged from 0 (no impairment) to 244 (maximum impairment), higher scores indicate increased impairment.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of the study drug. LOCF method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 208 | 206 | 208 | 206
units on a scale
  Baseline | 1.55 (3.45) | 1.75 (3.90) | 1.14 (3.32) | 1.43 (3.23)
  Change at Week 2 | -0.14 (1.34) | -0.37 (2.49) | 0.14 (2.28) | -0.20 (1.65)
  Change at Week 4 | -0.02 (1.78) | -0.50 (2.70) | -0.16 (2.20) | -0.25 (1.71)
  Change at Week 8 | -0.12 (2.14) | -0.51 (2.58) | -0.00 (2.71) | -0.27 (1.40)
  Change at Week 12 | -0.17 (1.88) | -0.42 (2.53) | -0.12 (2.67) | -0.25 (1.58)
  Change at Week 16 | -0.11 (1.70) | -0.50 (2.53) | -0.21 (2.69) | -0.34 (1.73)
  Change at Week 24 | -0.13 (1.75) | -0.51 (2.50) | -0.21 (2.69) | -0.34 (1.70)

38. Other Pre Specified Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA) Level
Description: Participants who developed anti-tanezumab antibodies after treatment were evaluated for the presence of anti-tanezumab neutralizing antibodies in their serum. Number of participants with positive ADA were summarized for reporting groups: tanezumab 5 mg + placebo and tanezumab 10 mg + placebo. Results with titer value >= 4.32 nanogram per milliliter of anti-tanezumab neutralizing antibodies were counted as positive.
Time Frame: Baseline, Week 8, 16, 24
Population: Analysis set included all randomized participants who received at least 1 dose of the study drug. This outcome measure was planned not to be analyzed for reporting arms: placebo and naproxen + placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo
Number analyzed (Participants) | 206 | 208
Participants
  Baseline | 1 | 1
  Week 8 | 1 | 0
  Week 16 | 0 | 0
  Week 24 | 1 | 1

39. Other Pre Specified Outcome: Number of Participants With Clinically Significant Changes in Vital Signs Abnormalities
Description: Assessment of the clinical significance of vital sign changes was done per investigator judgment. Changes in vital signs determined to be clinically significant by the investigator were reported as adverse events.
Time Frame: Day 1 (Baseline) up to Week 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 208 | 206 | 208 | 206
Participants | 2 | 0 | 2 | 3

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study. ITT analysis set evaluated for safety.
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Serious Adverse Events (participants affected / at risk) | 8/208 | 7/206 | 6/208 | 5/206
Other Adverse Events (participants affected / at risk) | 59/208 | 70/206 | 92/208 | 68/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=208) | Tanezumab 5 mg + Placebo (N=206) | Tanezumab 10 mg + Placebo (N=208) | Naproxen + Placebo (N=206)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Collapse of lung (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=208) | Tanezumab 5 mg + Placebo (N=206) | Tanezumab 10 mg + Placebo (N=208) | Naproxen + Placebo (N=206)
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 6
Nausea (Gastrointestinal disorders) | 4 | 4 | 4 | 6
Oedema peripheral (General disorders) | 0 | 9 | 15 | 4
Bronchitis (Infections and infestations) | 5 | 0 | 3 | 4
Influenza (Infections and infestations) | 4 | 0 | 5 | 3
Nasopharyngitis (Infections and infestations) | 4 | 2 | 6 | 8
Sinusitis (Infections and infestations) | 10 | 6 | 6 | 7
Upper respiratory tract infection (Infections and infestations) | 9 | 12 | 6 | 4
Urinary tract infection (Infections and infestations) | 2 | 6 | 7 | 7
Fall (Injury, poisoning and procedural complications) | 8 | 5 | 2 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 8 | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 12 | 14 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 3 | 7
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 7 | 8 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 4 | 5 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 6 | 20 | 1
Allodynia (Nervous system disorders) | 0 | 0 | 5 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 3 | 5 | 0
Dizziness (Nervous system disorders) | 5 | 6 | 0 | 3
Headache (Nervous system disorders) | 11 | 7 | 5 | 9
Hypoaesthesia (Nervous system disorders) | 2 | 4 | 10 | 7
Paraesthesia (Nervous system disorders) | 3 | 12 | 18 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction Description: Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.